CLINICAL TRIAL: NCT02101957
Title: Multicentric Trial of the Treatment of Huntington's Disease by Cysteamine (RP103)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHRC2004-03bis
Record Dates: First submitted 2014-03-25; First posted 2014-04-02 (Estimated); Last update posted 2014-04-02 (Estimated); Status verified 2013-07

CONDITIONS: Huntington's Disease
MeSH Terms: conditions — Huntington Disease

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- RP103 (Experimental): RP103 capsule, 16 capsules per day
  Interventions: Drug: RP103
- placebo (Placebo Comparator): placebo capsule, 16 capsules per day
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RP103
  Arms: RP103
Drug: Placebo
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the effect of cysteamine in patients with symptomatic Huntington's disease by comparing two groups of patients (cysteamine vs placebo) on the results of the Unified Huntington's Disease Rating Scale (UHDRS, Huntington study group 1996).

ELIGIBILITY:
Inclusion Criteria:

* Clinically disease-registered for at least one year, leading to consult (abnormal movements, neuropsychiatric disorders, neuropsychological impairment).
* Unified Huntington's Disease Rating Scale motor ≥ 5
* Total Functional Capacity > 10 (≥ 11)
* Huntington Disease diagnosed with abnormal number of CAG repeats: 38 < nucleotide expansion (CAG)
* Age between 18 and 65
* Voluntarily Patient Consent
* Patients willing and able to take oral medications, and comply with the specific procedures of the study

Exclusion Criteria:

* Severe cognitive impairment or neuropsychiatric troubles.
* No drug compliance to previous treatment.
* Patients with contra indication to the realization of imaging studies (including claustrophobia ) .
* Patients who have not given their written and informed consent signed .
* No national health insurance affiliation
* Private patients of their liberty by judicial or administrative decision, or patients under supervision.
* Pregnant women ( pregnancy test will be carried out systematically for women at risk) or lactating .
* Women who could become pregnant during the study period and with no contraception.
* Patients who have developed hypersensitivity to cysteamine or penicillamine ( against indication of cysteamine ) .
* Brain Damage intercurrent MRI. Brain morphological abnormalities , other than those characteristic of the disease .
* Disease - associated with neurological repercussions.
* Affection - visceral serious , scalable , involving life-threatening.
* Mental - disorder may disrupt accession to the Protocol , including a history of spontaneous and / or drug-induced hallucinations history of severe depression that required repeated hospitalizations , history of repeated suicide attempts .
* Participation in progress, or interrupted for less than three months, a therapeutic protocol of Huntington's disease .
* Patients with a history of surgical interventions to improve the symptoms of Huntington 's disease such as graft neuron, deep brain stimulation, infusion of neurotrophic agent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2010-10; Primary Completion 2015-07 (Estimated)

PRIMARY OUTCOMES:
Unified Huntington's Disease Rating Scale motor | at 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Angers, Angers, France